CLINICAL TRIAL: NCT03331705
Title: Evaluation of the Performance of a Disposable Cystoscope System for Direct Visualization of the Urethra and Bladder
Brief Title: Assessment of the Uro-C Cystoscope for Use in Diagnostic Cystoscopy Procedures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UroSee Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-001
Record Dates: First submitted 2017-10-26; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Bladder Tumor
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Use of new cystoscope: Patients in which the cystoscope is used.
  Interventions: Device: Uro-C (Use of new cystoscope)

INTERVENTIONS:
Device: Uro-C (Use of new cystoscope) — Diagnostic cystoscopic procedure of the urethra and bladder

SUMMARY:
This is a prospective, multicenter, single-arm, open-label clinical usability study in subjects who are candidates for office diagnostic cystoscopy. The primary objective of this initial device assessment is to evaluate the performance of a new cystoscope for direct visualization of the urethra and bladder.

DETAILED DESCRIPTION:
A new cystoscope has been designed for female diagnostic cystoscopy, with a focus on promoting patient comfort, tolerability and safety while improving office efficiency. The cystoscope, named the Uro-C, is light-weight, ergonomic, handheld, battery-operated portable system that integrates a disposable cannula with a reusable handle that contains video electronics, is wireless capable, and has a liquid crystal display (LCD) monitor. Cystoscopy with the new system is performed in a standard manner to cystoscopy with currently available endoscopes, so risks are no different than when currently available endoscopes are used.

This is a prospective, multi-center, single-arm, open-label clinical usability study in subjects who are candidates for office diagnostic cystoscopy. The primary objective of this initial device assessment is to evaluate the performance of the cystoscope for direct visualization of the urethra and bladder.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy adult (18 years of age or older) women presenting for cystoscopy for diagnostic purposes; and
2. Ambulatory and able to undergo routine cystoscopy in the lithotomy position.

Exclusion Criteria:

1. History of prior bladder/urethral surgery other than TURBT; or
2. History of interstitial cystitis; or
3. Presence of urinary tract infection (UTI); or
4. Gross hematuria; or
5. History of pelvic radiation therapy; or
6. Procidentia; or
7. Unable to read, understand, and/or provide a ranking of pain level during the procedure; or
8. Unable or unwilling to provide consent to participation in the study.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Females requiring a diagnostic cystoscopic procedure
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-11-05; Primary Completion 2018-07-05 (Estimated); Study Completion 2018-09-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of the utility and performance of the cystoscope by the physician | during the procedure
  Ranking with Likert Scale on ease of advancement, visibility of tissue and structures, and removal of the device

SECONDARY OUTCOMES:
Patient tolerance of the procedure | during and within 5 days after the procedure
  Assess level of discomfort or adverse event associated with the procedure by the subject using the Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Bela Denes, MD, Study Director — UroSee Corporation
Locations (1):
- Las Vegas Urology, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided